CLINICAL TRIAL: NCT01647841
Title: Maternal Determinants of HIV-exposed and HIV-unexposed Fetal Growth, Birth Outcomes and Early Infant Growth
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 1111002615
Record Dates: First submitted 2012-07-18; First posted 2012-07-24 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: HIV; Pregnancy; Malnutrition; Cachexia
MeSH Terms: conditions — Malnutrition; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women and infants: HIV+ and HIV- pregnant women, HIV-exposed and HIV-unexposed infants, ARV-exposed and ARV-unexposed infants

SUMMARY:
The purpose of this study is to understand how differences in the nutritional status and concentration of hormones and cytokines associated with cachexia in HIV+ and HIV- pregnant women living in a semi-rural and rural region of northern Tanzania affect fetal growth, pregnancy outcomes and early infant health and development. The study hypothesis is that HIV+ women will have worse nutritional status and a greater degree of cachexia which will negatively impact fetal growth, pregnancy outcomes and early infancy health and development.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by mothers, and parental consent on behalf of their infants
* Confirmed HIV status (HIV-1, HIV-2 or HIV-Dual seropositive or HIV-seronegative)
* Estimated gestational age between 12th and 34th weeks
* Stated intention to remain in the clinic catchment area ≥6 months post-partum
* Singleton birth

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: HIV+ and HIV- women and their infants attending a semi-rural clinic and/or rural dispensaries for their antenatal and early infancy care in north western Tanzania
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maternal cachexia score | Up to 1 month post-partum

SECONDARY OUTCOMES:
Maternal anthropometric measures | Up to 1 month post-partum
  weight, height, mid-upper arm circumference, triceps skinfold, fundal height
Fetal growth | Up to 1 month post-partum
Pregnancy outcomes | Up to 1 month post-partum
  spontaneous abortion, stillbirth, preterm delivery, perinatal mortality (death within first 7 days), neonatal mortality (death within first 28 days), small for gestational age, intrauterine growth retardation, low birth weight
Early infant anthropometrics | Up to 1 month post-partum
  weight, length, head circumference, mid-upper arm circumference, triceps skinfold

CONTACTS AND LOCATIONS:
Overall Officials: Joann M. McDermid, PhD, RD, Principal Investigator — Cornell University
Locations (1):
- Kisesa Health Centre, Kisesa, Tanzania